CLINICAL TRIAL: NCT04487093
Title: Clinical Study of Personalized Neoantigen Peptide Vaccine Combined With Targeted Drugs in the Treatment of Non-small Cell Lung Cancer
Brief Title: Clinical Study of Neoantigen Vaccine Combined With Targeted Drugs in the Treatment of Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Hospital of Shijiazhuang City (Other)
Collaborators: Tianjin Hengjia Biotechnology Development co., LTD (Industry)
Responsible Party: Principal Investigator, YAN ZHANG, Director of Oncology IV, First Hospital of Shijiazhuang City
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DYYY-2020-04-01
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non-small cell lung cancer; Individualized neoantigen peptides vaccine; Targeted Drugs; clinical trial; phase I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Patients enrolled without disease progression were given neoantigen vaccine combined with EGFR-TKI therapy； Patients with disease progression were given neoantigen vaccine combined with anti-angiogenesis drug therapy. Patients received subcutaneous injection of individualized neoantigen vaccines at a dose of 200ug per peptide once a week for 5 weeks. The targeted drugs are used continuously according to the instructions and dosage until disease progression or intolerance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoantigen vaccine + EGFR-TKI (Experimental)
  Interventions: Drug: neoantigen vaccine + EGFR-TKI
- neoantigen vaccine + anti-angioge (Experimental)
  Interventions: Drug: neoantigen vaccine + anti-angioge

INTERVENTIONS:
Drug: neoantigen vaccine + EGFR-TKI — Patients received subcutaneous injection of individualized neoantigen peptides vaccine at a dose of 200ug per peptide once a week for 5 weeks.
  The targeted drugs are used continuously according to the instructions and dosage until disease progression or intolerance.
  Arms: neoantigen vaccine + EGFR-TKI
Drug: neoantigen vaccine + anti-angioge — neoantigen vaccine + anti-angioge
  Arms: neoantigen vaccine + anti-angioge

SUMMARY:
Neoantigen vaccine is a new field of research in tumor immunotherapy, and some studies have been conducted with success on Melanoma and glioblastoma. Nearly 80% of lung cancers are diagnosed in an advanced stage (IIIB, and IV) and EGFR mutant non-small cell lung cancer will be resistant after targeted drug treatment. Neoantigen vaccine is a new treatment method for lung cancer, especially for patients with drug resistance.

DETAILED DESCRIPTION:
This is a phase I clinical study of individualized neoantigen peptide vaccine combined with targeted drugs in the treatment of EGFR mutant non-small cell lung cancer aimed to evaluated the safety and immune response of the neoantigen vaccine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced or metastatic non-small-cell lung cancer (stage III or stage IV).
2. With EGFR-TKI sensitive mutations and no T790M.
3. First generation EGFR-TKI treatment is in progress, the treatment time is 5-6 months and there is no disease progression.
4. Patients aged 18 to 85
5. Life expectancy of at least 3 months.
6. ECOG Performance Status 0 to 3.
7. No previous immunotherapy, including anti-PD-1/PD-L1 or co-suppressive T cell receptor drug therapy, peptide / mRNA neoantigen immunotherapy and cell therapy.
8. Ability to follow research and follow-up procedures. Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

1. Pregnant and/or breastfeeding.
2. With active, known or suspected autoimmune diseases or other concurrent immune system diseases.
3. Receive systemic cytotoxic chemotherapy or experimental drugs within 4 weeks before the start of neoantigen treatment, excluding EGFR-TKI and anti-angiogenesis targeted drugs.
4. Patients participated in other anticancer drug clinical trials within 4 weeks.
5. Liver and kidney dysfunction, severe heart disease, coagulation dysfunction, and impaired hematopoietic function.
6. Systemic infection.
7. Any uncertainties that have an impact on the safety or compliance of the patient.
8. Any disease, treatment, abnormal laboratory history or medical history that affects the participant's participation in the entire research process, or the investigator believes that it is not suitable to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-17 (Actual); Primary Completion 2022-05-17 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03. | 24 months
  Safety

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 2 years
  PFS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Overall survival (OS) | Up to 2 years
  OS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Disease Control Rate(DCR) | Up to 12 weeks
  DCR as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M.D., Study Chair — The First Hospital of Shijiazhuang
Locations (1):
- The First Hospital of Shijiazhuang, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No